CLINICAL TRIAL: NCT01268345
Title: AST Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andon Medical Co.,Ltd (Industry)
Responsible Party: Yi Liu, Andon Medical Co.,Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AndonMedical2
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes
Keywords: blood glucose
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Andon (Experimental): Andon blood glucose test strips with test meter
  Interventions: Device: blood glucose monitor
- Lifescan (Active Comparator)
  Interventions: Device: blood glucose monitor

INTERVENTIONS:
Device: blood glucose monitor — Blood glucose monitor is used to monitor the blood glucose level of the human-being
  Other Names: Andon blood glucose monitor
  Arms: Andon
Device: blood glucose monitor — Blood glucose monitor is used to monitor the blood glucose level of the human-being.
  Other Names: Lifescan blood glucose monitor
  Arms: Lifescan

SUMMARY:
Blood glucose monitoring system are tested in the alternative site to validate the accuracy of the blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* people ( disbetes people)with at least 8 hours of limosis

Exclusion Criteria:

* After meal(when doing the test)
* take Hypoglycemic Drugs(when doing the test)
* with insulin(when doing the test)
* after strenuous exercise(when doing the test)
* Pregnant women
* neonates
* patients in a hyperglycemic-hyperosmolur state, with or without ketosis.
* patients who are dehydrated, hypertensive, hypotensive or in shock.

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
blood glucose value | 5 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Hexi Ruijing metabolism hospital, Tianjin, Tianjin Municipality, China